CLINICAL TRIAL: NCT05355038
Title: Effect of Lifestyle Modification on Pregnancy Outcomes for Pregnant Women With Gestational Diabetes: an Evidence Based.
Brief Title: Effect of Lifestyle Modification on Pregnancy Outcome for GDM
Acronym: Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Said Mahmoud Elgamasy, assistant lecture in maternal and newborn health nursing, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Basma said Mahmoud El gamasy
Record Dates: First submitted 2022-04-02; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: GDM; Lifestyle; Pregnancy Outcome
MeSH Terms: interventions — Diet Therapy; Exercise; Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: control and study group
Who Masked: Participant
Masking Description: control group were in the first 3 day of week (saturday ,sunday ,monday) study group were in the 2nd three day of week(tuesday, wednsday,thursday)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lifesyle modification (Experimental): intervention group will take lifestyle modification protocol which composed of health teaching about low glycemic index diet, physical activity and self glucose monitoring
  Interventions: Behavioral: lifestyle modification (dietary modification); Behavioral: lifestyle modification (physical activity); Behavioral: lifestyle modification( self glucose monitoring)
- control group (No Intervention): routine care of the hospital

INTERVENTIONS:
Behavioral: lifestyle modification (dietary modification) — low glycemic index diet the researcher gave detail information about (importance of LGI diet, component of food, number of meals and snake, example of food taken in breakfast, lunch, dinner and snake in between, food allowed and not allowed). After that, the researcher required from the woman to make an example of food for one day according to her income level, if correction of the content of food needed, the researcher will explain this point again.
  Other Names: low glycemic index diet
  Arms: lifesyle modification
Behavioral: lifestyle modification (physical activity) — health teaching about choose between two types of exercise to be selected according to the ability of GDM women to perform : brisk walking or seated arm exercise or selected both. Brisk walking should be performed for at least half an hour three time /week, while, seated arm exercise done three time after each meal for10 minute in each time. The researcher given a detail information about both types and its importance in decreasing blood glucose level, also how to perform and what should be done in case of appearance of fatigue manifestation during exercise, and the women have choice for perform both or selected one to perform according to your health condition.
  Other Names: brisk waking exercise or seated arm exercise or both type performed
  Arms: lifesyle modification
Behavioral: lifestyle modification( self glucose monitoring) — self-glucose monitoring the researcher explain the important of monitoring blood glucose level and instruct the women about how to perform self- glucose measuring, recording way of the result in schedule and to bring this result in the next antenatal visit. The women who have digital blood glucose monitoring instructed to measure it at least 5 time/day. while, the women who didn't have digital blood glucose monitoring measure went to nearest pharmacy to measure blood glucose at least one time per day especially when the woman felt the signs and symptoms of hypo or hyperglycemia and recorded the result in paper or sent the result in whatsapp for the researcher if you have whatsapp application. In addition to give the woman instruction about sings symptoms of hypoglycemia and hyperglycemia and the proper ways for management
  Other Names: self glucose monitoring
  Arms: lifesyle modification

SUMMARY:
Effect of lifestyle modification on pregnancy outcome for pregnant women with GDM

DETAILED DESCRIPTION:
evaluate the effect of lifestyle modification on pregnancy outcome among GDM women.

Primary outcomes: excessive gestational weight gain, uncontrolled blood glucose level, PIH, polyhydromnios, oligohydrominos, recurrent monilia infection and urinary tract infection , intra uterine fetal death (IUFD), intra uterine growth restriction (IUGR), premature preterm rupture of membrane and Diabetic ketoacidosis.

Secondary outcomes: preterm labor, caesarian section, neonatal hypoglycemia, stillbirth, respiratory distress syndrome, small for gestational age (SGA), large for gestational age (LGA) ,neonatal intensive care unit (NICU) and failure to initiate or maintain breast feeding.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with GDM

Exclusion Criteria:

* pre-gestational diabetes type 1 or type 2 diabetes mellitus, diagnosed as pregnancy induced hypertension before GDM

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  change blood glucose level (fasting blood sugar (FBS) and random blood sugar (RBS) measured with digital blood glucose monitoring by using test strips; HA1C and urine analysis done in the laboratory and get the result)
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  attained proper weight gain during pregnancy. Weight was measured utilizing bath scale where the accuracy were obtained through balancing zero prior weighting
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  occurrence of maternal complications during pregnancy((preeclampsia, urinary infection, monilia infection, premature rupture of membrane, bleeding during pregnancy, and diabetic ketoacidosis).this will recorded by using tool to assess this compilication
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  occurrences of fetal complications during pregnancy detected by the result of ultrasound done by physician (decrease fetal movement count, IUGR, and IUFD)
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  Intrapartum assessment of the outcomes. The researcher assessed mode of delivery and complications occurrence to the GDM women and their neonatal during intrapartum from the hospital filling . The maternal complications (preterm labor, prolonged labor, traumatic labor, intrapartum instrumental delivery, perineal trauma or tear, postoperative hemorrhage and infection). While regarding to fetal assessment (occurrences of intra uterine fetal death, preterm birth, Birth trauma (shoulder dystocia, bone fracture, cerebral palsy), fetal distress, macrosomia, IUGR, five-minute Apgar less than seven, stillbirth)
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  Postpartum assessment of the outcomes.The researcher assessed each woman and their newborn for the first 24 hours postpartum in both groups. It included the following items:1) assessed maternal vital sings: Temperature was assessed by using thermometer; blood pressure was measured through a sphygmomanometer; 2) maternal and newborn lab investigation as FBS and postprandial using digital blood glucose monitoring with test strips.
  In addition to, assess the occurrences of Maternal and newborn complications as; postpartum hemorrhage, failure or delay for initiating breastfeeding, neonatal hypoglycemia, respiratory distress syndrome, sings of jaundice, (SGA or LGA), neonatal death, and neonatal administration to ICU, and preterm birth.
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  newborn gestational age. assessment of the neonatal anthropometric measurements such as weight which taken from labor sheet, length was measured from head to toe when the neonates were in supine position and legs were extended using measurement tap. Then, measured head circumference through measurement tape firmly around head above the eyebrow ridge. The researcher plotted neonatal weight, length and head circumference by gestational age on the growth chart, to determine if the growth below 10th percentile the neonate was small for gestational age (SGA), if the growth above the 90th percentile, the neonates was large for gestational age (LGA) called macrocosmic baby, if the growth was in between 10th and 90th percentiles, the neonates was appropriate for gestational age (AGA). Postpartum assessment taken 30 minutes for each woman in each group.
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  body mass index(was calculated through the formula "weight in Kg, divided by height squared in meters"; class of weight using the international classification of adult underweight<18.5, normal weight 18.5-24.9, over weight 25-29.9 and obesity ≥ 30 according to BMI )
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  height measured by using measurement tape. firstStand with your feet flat on the floor with your heels against the corner where the wall and floor meet. Make sure your head, shoulders, and buttocks are touching the wall. then use Use a tape measure - - to measure the distance from the floor to the mark on the wall.
  Stand up straight with your eyes looking straight ahead. Your line of sight and chin should be parallel to the floor.
effect of lifestyle modification among GDM on pregnancy outcome | from 28 weeks of gestational until the first 24hours postpartum
  assessment of fasting blood sugar and random blood sugar for the postpartum GDM women and their neonatal in the first 24 hours postpartum by using (fasting blood sugar (FBS) and random blood sugar (RBS) measured with digital blood glucose monitoring by using test strips

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Cairo, Egypt